CLINICAL TRIAL: NCT01604174
Title: Effectiveness of an Interactive Virtual Telerehabilitation System in Patients After Total Knee Arthroplasty. A Randomized Controlled Trial
Brief Title: Interactive Virtual Telerehabilitation After Total Knee Arthroplasty
Acronym: REHABITIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REHABITIC
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; arthroplasty; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Virtual Telerehabilitation (Experimental): Rehabilitation by IVT
  Interventions: Other: Interactive Virtual Telerehabilitation (IVT)
- Standard rehabilitation care (Active Comparator): Standard care rehabilitation after total knee arthroplasty
  Interventions: Other: Standard care rehabilitation

INTERVENTIONS:
Other: Interactive Virtual Telerehabilitation (IVT) — Rehabilitation after arthroplasty of knee using IVT
  Other Names: Rehabilitation procedure (physical manipulation) plus IVT
  Arms: Interactive Virtual Telerehabilitation
Other: Standard care rehabilitation — Standard care rehabilitation after total knee arthroplasty
  Other Names: Rehabilitation procedure (physical manipulation)
  Arms: Standard rehabilitation care

SUMMARY:
The purpose of this clinical trial is to compare the effectiveness of a new interactive virtual telerehabilitation (IVT) system with the conventional program in the rehabilitation of patients after total knee arthroplasty.

DETAILED DESCRIPTION:
Patients are distributed into two treatment groups: 1) Group I (control): standard clinical protocol of TKA rehabilitation consisting of 1-hour sessions for 10 days; and 2) Group II (IVT): 1-hour IVT sessions for 10 days (5 sessions under a therapist's supervision to verify the absence of medical complications + 5 sessions performed at home). The IVT is an interactive virtual software-hardware platform that facilitates the development of remote rehabilitation therapy for multiple diseases. Patients receive information required to perform exercise and the therapist remotely monitors the patient's performance. For the purpose of this trial, the IVT system was designed for lower limb motor recovery in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Post-TKA active range of motion: flexion 80º and extension -10º
* ABsence of stiffness
* Ability to walk with the use of a walking aid
* Ability to read and understand Spanish
* Ability to understand and accept the trial procedures and to sign an informed consent form in accordance with national legislation

Exclusion Criteria:

* Sensory, cognitive and/or praxic impairment
* Concomitant medical conditions that may influence the rehabilitation process
* Discharge destination other than home
* Patients with any local or systemic complication (e.g., surgical wound infection, suspicion of deep vein thrombosis…) in the three-month follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Active knee extension/flexion | Change from baseline to 2 weeks
  Active knee extension/flexion measured by investigator

SECONDARY OUTCOMES:
Muscle strength | Baseline to 2 weeks
  Measure of muscle stregth by investigator. That include measures of strength of the quadriceps, Harmstring muscle strength and Timed Getr-UP-ang-Go test
Pain | Baseline to 2 weeks
  Measure of pain by visual analog scales
Functional capacity | Baseline to 2 weeks
  Measure of functional capacity using questionnaires /Western Ontario and MacMaster University)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Muniesa, MD, PhD, Principal Investigator — Parc de Salut Mar; Ferran Escalada, Md, PhD, Study Director — Parc de Salut Mar
Locations (1):
- Hospital del Mar (PSMAR), Barcelona, Barcelona, Spain